## "The effects of Neurodevelopmental Therapy on Feeding and Swallowing Activities in Children with Cerebral Palsy"

NCT04403113

27.03.2018

## **Informed Consent Form**

I would like to do research called "The Evaluation of the Effect of Trunk Stabilization Exercises on Feeding and Swallowing Activity in Children with Cerebral Palsy". This research will evaluate how your child performs an eating activity and uses trunk muscles. The research will be performed under the direction of Assoc. Dr Gönül ACAR, and Pt. Nasim EJRAEI from Marmara University Health Sciences Institute, Department of Physiotherapy and Rehabilitation.

You are invited to a study. It is very important to understand why and how to research before making a decision. Please take some time and carefully read the information below, discuss with others if you wish. If there is an unclear section or if you need more detailed information, you can get information from us. But please consider a little bit to decide if you want to participate in the research. You are invited to our research because you meet the criteria for inclusion in the research sought by the participants. Children who volunteer to participate in this study will either receive oral-motor therapy in addition to the physiotherapy program applied based on the principles the Neurodevelopmental Treatment or will receive therapy that includes trunk exercises in addition to physiotherapy and oral-motor therapy. Both types of therapy programs do not harm your child without any special risks. Before and after this exercise program, your child will be evaluated.

We would like to point out that participation is voluntary and refusal to participate will not lead to any punishment or loss of any benefit. Likewise, after you agree to participate in the research, you can withdraw from the research without showing any reason anywhere in the research.

The assessments applied to the participants participating in our research have no known harm. In case of any unexpected loss arising during the evaluation process, the information will be given immediately. If you are harmed in any way from the evaluations, the necessary applications will be met by the researchers without any response. No fees will be charged for this, neither from you nor from your Social Security.

Although it may be beneficial for you to participate in the research immediately, it is hoped that our research results will benefit the institution, society or science in the future.

I have read the entire information form clearly or understandably read/translated to me as

I do not know the language/reading. I was allowed to ask, evaluate and make decisions about

my health status both during and after my application and while filling out this form. All

treatment and diagnostic alternatives, including the possibility of non-treatment, and whether

there are risks and dangers were explained.

Name-Surname of the participant and his/her legal representative:

**Date/Signature:** 

I gave the patient the necessary information about the disease and the procedures to be

applied. I believe that the patient understands this information, asks me the questions he wants

to ask, and accepts the process with his free will.

Researcher: Pt. Nasim EJRAEI

Address: Marmara University Başıbüyük Health Campus, Health Sciences Institute

Directorate, Başıbüyük Yolu 9/3 34854 Başıbüyük/ Maltepe/ Istanbul

**Telephone:** 0539 298 71 26

**E-mail:** ejraeinasim@yahoo.com

**Date/Signature:**